CLINICAL TRIAL: NCT06682637
Title: Melflufen for Elderly Myeloma Patients in Second or Subsequent Relapse
Brief Title: Melflufen for Elderly Patients With Relapsed Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical trial never activated, not authorized by CA
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MELISSA
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Relapse Multiple Myeloma
MeSH Terms: interventions — melflufen; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Treatment consists in 28-day cycles:
  * Melflufen 40 mg total dose (30 mg in patients with body weight ≤60 kg and/or in patients with eGFR<45 mL/min) intravenously on day 1.
  * Dexamethasone 10 mg orally or intravenously on day 1-2, 8-9, 15-16, 22-23. Cycles are repeated until clinical relapse or progression, or unacceptable toxicity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Melflufen and Dexamethasone (Experimental): * Melflufen 40 mg total dose (30 mg in patients with body weight ≤60 kg and/or in patients with eGFR<45 mL/min) intravenously on day 1.
  * Dexamethasone 10 mg orally or intravenously on day 1-2, 8-9, 15-16, 22-23.
  Interventions: Drug: Melflufen; Drug: Dexamethasone

INTERVENTIONS:
Drug: Melflufen — Pepaxti 20 mg powder for concentrate for solution for infusion
Drug: Dexamethasone — SOLDESAM 8 mg/2 ml solution for injection SOLDESAM 0.2% oral drops, solution

SUMMARY:
This is a pilot study aimed to evaluate the efficacy and tolerability of melflufen plus dexamethasone in elderly patients at second relapse.

Thirty elderly patients at second or subsequent relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by MM progressed or relapsed after 2 or more previous lines of therapy.
* Patient is, in the investigator's opinion, willing and able to comply with the study visits and procedures required per protocol.
* Patient has provided written informed consent in accordance with federal, local, and institutional guidelines prior to initiation of any study-specific activities or procedures. Subject does not have kind of condition that, in the opinion of the Investigator, may compromise the ability of the subject to give written informed consent and patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Life expectancy ≥ 3 months
* Previous exposure to, at least, one drug of all the following categories: an anti-CD38 MoAbs, an IMiD, and a proteasome inhibitor.
* Age ≥ 70 and ≤ 85 years.
* ECOG performance status ≤2.
* Subject must have serum monoclonal paraprotein (M-protein) level ≥0.5 g/dL or urine M-protein level ≥200 mg/24 hours, or serum immunoglobulin involved free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio.
* LVEF ≥40% as determined by a MUGA scan or ECHO.
* Adequate hepatic function characterized by the following:

oTotal bilirubin ≤1.5 x ULN. oAST ≤2.5 x ULN oALT ≤2.5 x ULN.

* Estimated creatinine clearance ≥30 mL/min (according to the Cockcroft Gault formula, by 24-hour urine collection for creatinine clearance, or per the local institutional standard method).
* Adequate BM function characterized by the following:

  * Absolute neutrophil count ≥1.0 × 109/L (use of granulocyte-colony stimulating factors is permitted if completed at least 7 days prior to planned start of dosing).
  * Platelet count ≥50 × 109/L (transfusion support is not permitted).
  * Hemoglobin ≥8 g/dL (transfusion support is permitted).
* Non-vasectomized male patients agree to practice appropriate methods of birth control

Exclusion Criteria:

* Previous exposure to chemotherapy (i.e. melphalan, high-dose melphalan and/or cyclophosphamide) with the exception of patients who have received an autologous stem cell transplantion with a progression free survival of at least 36 month.
* Plasma cell leukemia.
* Systemic amyloid light chain amyloidosis.
* POEMS Syndrome.
* Central Nervous System (CNS) disease localization.
* Subject with another tumor, not including MM, that required ongoing treatment or therapy completed less than 6 months before eligibility confirmation, and considered at substantial risk of relapse in the following 12 months.
* Active HBV, HCV, SARS-CoV2, HIV, or any active, uncontrolled bacterial, fungal, or viral infection. Active infections must be resolved at least 14 days prior to eligibility confirmation.
* Subject has any concurrent medical condition or disease (e.g. active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
* Subject has clinically significant cardiac disease, including:

  * Myocardial infarction within 6 months before trial eligibility
  * Uncontrolled disease/condition related to or affecting cardiac function (e.g. unstable angina, congestive heart failure, New York Heart Association Class III-IV)
  * Clinically significant ECG abnormalities.

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | approximately 6 months after the enrolled of the last participant and an updated analysis will be conducted at approximately 8 to 12 months.
  rate of participants who achieve a PR or better (PR+VGPR+CR+sCR) according to IMWG response criteria during the treatment.

SECONDARY OUTCOMES:
DURATION OF RESPONSE | after 2.5 years
  the time from the date of first documented response (≥PR) to the date of first confirmed PD.
PROGRESSION-FREE SURVIVAL | after 6 months
  the time from the date of 1st dose of study drug to the date of first confirmed PD or death due to any cause, whichever occurs first.
TIME TO PROGRESSION | after 2.5 years
  the time from the date of 1st dose of study drug to the date of first documented PD
PROGRESSION-FREE SURVIVAL 2 | after 2.5 years
  the time from the date of 1st dose of study drug to the date of event, which is defined as death from any cause or PD that starts after the next line of therapy, whichever occurs first.
OVERALL SURVIVAL | after 2.5 years
  the time from the date of 1st dose of study drug to the date of death.
TIME TO RESPONSE | after 2.5 years
  the time from the date of 1st dose of study drug to the first documented response (≥PR).

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - A.O.U. delle Marche, Ancona
  - Ospedale Nuovo di Legnano, Legnano
  - Ospedale Niguarda, Milan
  - Ospedale S. Carlo Borromeo, Milan
  - Policlinico Giaccone Divisione Ematologia e Centro Trapianti di Midollo, Palermo
  - A.O.U. di Parma, Parma
  - A.O.U. Pisana, Pisa
  - I.R.C.C.S. Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - A.O.U. Città della Salute e della Scienza di Torino-SSD Clinical trials, Torino
  - Ospedale S. Maria della Misericordia di Udine, Udine

IPD SHARING:
Plan to Share IPD: No